CLINICAL TRIAL: NCT01805622
Title: Efficacy to Effectiveness Transition of an Educational Program to Increase Colorectal Cancer Screening
Brief Title: Educational Program to Increase Colorectal Cancer Screening: a Cluster Trial
Acronym: EPICS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Morehouse School of Medicine (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Selina A. Smith, Principal Investigator, Morehouse School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: EPICS cRCT; 1R01CA166785 (NIH)
Record Dates: First submitted 2013-03-01; First posted 2013-03-06 (Estimated); Last update posted 2013-03-06 (Estimated); Status verified 2013-03

CONDITIONS: Colorectal Cancer
Keywords: community-based participatory research; colorectal cancer screening
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Passive Arm #1 (Experimental): Active Arm #1, 2; Passive Arm #1, 2 Community coalitions randomized to the Passive Arm #1-Web Access Without Technical Assistance will receive access to EPICS facilitator training materials and toolkits via the Research-Tested Intervention Programs (RTIPs) website and will not participate in monthly technical assistance teleconferences.
  Interventions: Behavioral: Active Arm #1, #2, Passive Arm #1, #2
- Passive Arm #2 (Experimental): Active Arm #1, #2; Passive Arm #1, #2 Community coalitions randomized to the Passive Arm #2-Web Access With Technical Assistance will receive access to EPICS facilitator training materials and toolkits via the Research-Tested Intervention Programs (RTIPs) website and will participate in monthly technical assistance teleconferences.
  Interventions: Behavioral: Active Arm #1, #2, Passive Arm #1, #2
- Active Arm #1 (Active Comparator): Active Arm #1, #2; Passive Arm #1, #2 Community coalitions randomized to Active Arm #1-In-Person Access Without Technical Assistance will receive training from intervention developers with access to facilitator training materials but will not participate in monthly technical assistance teleconferences.
  Interventions: Behavioral: Active Arm #1, #2, Passive Arm #1, #2
- Active Arm #2 (Active Comparator): Active Arm #1, #2; Passive Arm #1, #2 Community coalitions randomized to Active Arm #2-In-Person Access with Technical Assistance will receive training from intervention developers with access to facilitator training materials and will participate in monthly technical assistance teleconferences.
  Interventions: Behavioral: Active Arm #1, #2, Passive Arm #1, #2

INTERVENTIONS:
Behavioral: Active Arm #1, #2, Passive Arm #1, #2 — This four-arm cluster randomized trial (five community coalitions plus 1,800 African Americans, 50-74 years of age, who are not current on CRC screening per arm) compares the following implementation strategies: (1) web access to facilitator training materials and toolkits without technical assistance (TA); (2) web access, but with technical assistance (TA); (3) in-person access to facilitator training materials and toolkits without TA and (4) in-person access with TA.

SUMMARY:
* Hypothesis 1. When compared to passive dissemination, active dissemination will result in greater participant enrollment.
* Hypothesis 2. The intervention will be offered with equal fidelity in churches, clinics and community sites.
* Hypothesis 3. Knowledge of CRC screening and perceived risk of CRC will be positively correlated.

DETAILED DESCRIPTION:
In this study, investigators aim to evaluate 20 community coalitions and 7,200 participants by: testing passive and active approaches to disseminating the Educational Program to Increase Colorectal Cancer Screening (EPICS) to increase screening rates for colorectal cancer; measuring the extent to which EPICS is accepted and the fidelity of implementation in various settings and estimating the potential translatability and public health impact of EPICS. This four-arm cluster randomized trial (five community coalitions plus 1,800 African Americans, 50-74 years of age, who are not current on colorectal cancer (CRC) screening per arm) compares the following implementation strategies: (1) web access to facilitator training materials and toolkits without technical assistance (TA); (2) web access, but with technical assistance (TA); (3) in-person access to facilitator training materials and toolkits without TA and (4) in-person access with TA. Primary outcome measures are the reach (the proportion of representative eligible community coalitions and individuals participating in the trial) and effectiveness (post-intervention changes in CRC screening rates). Secondary outcomes include adoption (percentage of community coalitions implementing the EPICS sessions) and implementation (quality and consistency of the intervention delivery). The extent to which community coalitions continue to implement EPICS post-implementation (maintenance) will also be measured. Cost-effectiveness analysis will be conducted to compare passive to active dissemination costs. Investigators believe that implementing this evidence-based colorectal cancer screening intervention in partnership with community coalitions will result in more rapid adoption than traditional top-down approaches, and that changes in community CRC screening practices are more likely to be sustainable over time. With its national reach, this study has the potential to enhance understanding of barriers and enablers to the uptake of educational programs aimed at eliminating cancer health disparities.

ELIGIBILITY:
Inclusion Criteria:

* African Americans, 50-74 years of age, who are not current on CRC screening, are eligible for study participation

Exclusion Criteria:

* Individuals with a personal history of CRC or inflammatory bowel disease, blindness or severe hearing impairment; dementia; or other condition with life expectancy less than two years, are ineligible for participation

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7200 (Estimated)
Dates: Start 2012-08; Primary Completion 2017-03 (Estimated); Study Completion 2017-03 (Estimated)

PRIMARY OUTCOMES:
Reach (RE-AIM Framework) | up to 12 months
  The proportion of representative eligible community coalitions and individuals participating in the trial.
Effectiveness (RE-AIM Framework) | up to 24 months
  Post-intervention changes in CRC screening rates.

SECONDARY OUTCOMES:
Adoption (RE-AIM Framework) | up to 36 months
  Percentage of community coalitions implementing the EPICS sessions.
Implementation (RE-AIM Framework) | up to 36 months
  Quality and consistency of the intervention delivery.

OTHER OUTCOMES:
Maintenance (RE-AIM Framework) | up to 24 months
  The extent to which community coalitions continue to implement EPICS post-implementation.
Cost-effectiveness analysis | up to 60 months
  Compare passive to active dissemination costs.

CONTACTS AND LOCATIONS:
Overall Officials: Selina A. Smith, PhD, MDiv, Principal Investigator — Morehouse School of Medicine; Daniel S. Blumenthal, MD, MPH, Principal Investigator — Morehouse School of Medicine
Locations (1):
- Morehouse School of Medicine, Atlanta, Georgia, United States

REFERENCES:
- [Background] Smith S, Johnson L, Wesley D, Turner KB, McCray G, Sheats J, Blumenthal D. Translation to practice of an intervention to promote colorectal cancer screening among African Americans. Clin Transl Sci. 2012 Oct;5(5):412-5. doi: 10.1111/j.1752-8062.2012.00439.x. Epub 2012 Aug 7. PMID 23067354
- [Background] Smith SA, Blumenthal DS. Community health workers support community-based participatory research ethics: lessons learned along the research-to-practice-to-community continuum. J Health Care Poor Underserved. 2012 Nov;23(4 Suppl):77-87. doi: 10.1353/hpu.2012.0156. PMID 23124502
- [Derived] Ansa BE, Alema-Mensah E, Sheats JQ, Mubasher M, Akintobi TH. Colorectal Cancer Knowledge and Screening Change in African Americans: Implementation Phase Results of the EPICS Cluster RCT. AJPM Focus. 2023 Jun 13;2(4):100121. doi: 10.1016/j.focus.2023.100121. eCollection 2023 Dec. PMID 37790949
- [Derived] Smith SA, Blumenthal DS. Efficacy to effectiveness transition of an Educational Program to Increase Colorectal Cancer Screening (EPICS): study protocol of a cluster randomized controlled trial. Implement Sci. 2013 Aug 7;8:86. doi: 10.1186/1748-5908-8-86. PMID 23924263